CLINICAL TRIAL: NCT00877084
Title: Exacerbation and Training - Study; a Randomized Controlled Study of the Effect of Resistance Training in Acute Exacerbations of COPD
Brief Title: Exacerbation and Training in Patients With Chronic Obstructive Pulmonary Disease
Acronym: EXTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Fonds voor Wetenschappelijk Onderzoek-Vlaanderen, Research Foundation Flanders
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.5.139.06KAN
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: COPD
Keywords: exacerbation; COPD; Resistance training; Muscle force
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Resistance training: series of 3x8 repetitions will be performed for the quadriceps muscle at 70% of the 1 Repetition Maximum determined as the weight the patient can lift once over the full range of motion. The weight can be applied using free weights or using a classical multi-gym device or a quadriceps chair.
  Interventions: Other: Resistance training
- 2 (Placebo Comparator): Usual care according to clinical pathway for COPD exacerbations + NO training
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Resistance training — Resistance training: series of 3x8 repetitions will be performed for the quadriceps muscle at 70% of the 1 Repetition Maximum determined as the weight the patient can lift once over the full range of motion. The weight can be applied using free weights or using a classical multi-gym device or a quadriceps chair.
  Other Names: Usual care according to a clinical pathway + Resistance training
  Arms: 1
Other: Usual care — usual care according to clinical pathway for COPD, No training
  Arms: 2

SUMMARY:
When patients with chronic obstructive lung disease (COPD) are admitted to the hospital with a severe exacerbation they lose muscle strength. This muscle weakness predisposes these patients to further hospital admissions. Resistance training is a potent countermeasure to prevent and treat muscle weakness. In the setting of an acute exacerbation this intervention however has not been validated.

The present study aims at investigating the safety and efficacy of resistance training (3x8 quadriceps extensions per day) to prevent muscle weakness. End points are quadriceps muscle strength and hospital readmission and functional status at discharge. Using the minimally invasive needle muscle biopsy technique described by Bergström the effects of resistance training on the skeletal muscle will be analyzed in detail.

After giving informed consent, patients will be randomized on admission into usual care or usual care plus resistance training. Patients will be followed-up using the clinical pathway for COPD (10 days). After one month patients will attend the outpatient clinic for a follow-up visit. Besides the measurement prescribed in the clinical path for COPD (including arterial blood gas measures, lung function, functional investigation of the patients), patients will undergo muscle strength measures and venous blood will be drawn for the analysis of systemic inflammatory and growth factors. Half of the patients will receive a resistance training program. At the end of the hospital admission, a needle biopsy of the vastus lateralis muscle will be obtained.

ELIGIBILITY:
Inclusion criteria:

* COPD exacerbation, admitted to the respiratory units
* Informed consent
* Age < 80
* No critical comorbidity compromising outcome up to one month.
* No suspect of malignancy

Exclusion criteria:

* Patient is involved in a rehabilitation program with a frequency >1/wk during one month after inclusion in the study
* NIMV or ICU on admission
* Patient scheduled for procedure (LTX/LVRS) within one month after discharge
* Readmission <14 days after previous hospitalization
* Significant pathology that would hinder the participation in resistance training (gonarthrosis, arthritis to be judged by the investigator)
* Clinical signs of pulmonary hypertension

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-01; Primary Completion 2005-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Reduction in the decline of muscle force during the exacerbation. | discharge Day 9

SECONDARY OUTCOMES:
Time to readmission or death | 6 Months
Functional exercise capacity at discharge (6MWT) | discharge Day 9
Functional exercise capacity and muscle force at 1 month | 1 Month
Markers of systemic inflammation and oxidative stress in serum and muscle of patients at day 9 of the exacerbation. | Day 9

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Leuven, Campus Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Derived] Troosters T, Probst VS, Crul T, Pitta F, Gayan-Ramirez G, Decramer M, Gosselink R. Resistance training prevents deterioration in quadriceps muscle function during acute exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2010 May 15;181(10):1072-7. doi: 10.1164/rccm.200908-1203OC. Epub 2010 Feb 4. PMID 20133927